CLINICAL TRIAL: NCT03513484
Title: Phase Ib, Open Label, Combination Study of Nintedanib With 5-Azacitidine in Acute Myeloid Leukemia Characterized by HOX Gene Overexpression, That Are Not Candidates of Intensive Chemotherapy
Brief Title: Nintedanib and Azacitidine in Treating Participants With HOX Gene Overexpression Relapsed or Refractory Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Robert H. Lurie Cancer Center (Other); Boehringer Ingelheim (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 17H04; NCI-2018-00483 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00206525; NU 17H04 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia With t(9;11)(p22.3;q23.3); MLLT3-KMT2A; Fibroblast Growth Factor Basic Form Measurement; FLT3 Internal Tandem Duplication; Recurrent Adult Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (nintedanib, azacitidine) (Experimental): Participants receive nintedanib PO BID on days 1-28 and azacitidine IV or SC on days 1-7. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 courses, participants may discontinue treatment, receive nintedanib every 4-8 weeks, or receive nintedanib and azacitidine every 4-8 weeks.
  Interventions: Drug: Azacitidine; Other: Laboratory Biomarker Analysis; Drug: Nintedanib

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nintedanib — Given PO
  Other Names: BIBF 1120; BIBF-1120; Intedanib; Multitargeted Tyrosine Kinase Inhibitor BIBF 1120; tyrosine kinase inhibitor BIBF 1120; Vargatef

SUMMARY:
The purpose of this study is to find the appropriate dose of the study drug nintedanib when combined with azacitidine and the associated side effects of the combination in older adults with AML characterized by HOX gene overexpression who are not interested in or not considered fit for standard intensive chemotherapy. The use of the study drug nintedanib in this study is investigational. Investigational means that this medication has not yet been approved by the FDA to treat this type of cancer. Azacitidine received FDA Approval in 2004 for myelodysplastic syndrome (a blood cancer related to AML) and has a National Comprehensive Cancer Network (NCCN) guideline recommendation for treatment of older adults who are not candidates for or decline intensive remission induction therapy. We expect participation to continue in this study based on each participant's response to the drug, and ability to tolerate treatment. Participants may continue to receive study treatments for 6 cycles (one cycle is 28 days long). If the 6 cycles of treatment is completed, participants may be moved on to a maintenance phase of treatment. Treatment will continue until the participant's leukemia gets worse, or they experience serious side effects, have a break in treatment for more than 56 days or the study doctor feels it is best for study treatments to stop.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify maximum tolerated dose (MTD) of nintedanib for combination treatment of nintedanib and azacytidine (5-azacitidine) in the treatment of newly diagnosed and relapsed/refractory acute myeloid leukemia with HOX overexpression and who are ineligible for intensive chemotherapy.

SECONDARY OBJECTIVES:

I. Adverse events (AEs) including dose limiting toxicities (DLTs) will be assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 4.03.

II. To determine median overall survival. III. To determine complete remission (CR) rate.

EXPLORATORY OBJECTIVES:

I. To determine composite CR rate (CR + complete remission with incomplete platelet recovery [CRp] + complete remission with incomplete hematological recovery [Cri]).

II. To determine duration of confirmed response. III. To determine event free survival. IV. To determine leukemia free survival. V. To establish correlation between response and pre-treatment Fgf2 levels and change in Fgf-2 levels during treatment.

OUTLINE: This is a dose-escalation study of azacitidine.

Participants receive nintedanib orally (PO) twice daily (BID) on days 1-28 and azacitidine intravenously (IV) or subcutaneously (SC) on days 1-7. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 courses, participants may discontinue treatment, receive nintedanib every 4-8 weeks, or receive nintedanib and azacitidine every 4-8 weeks.

After completion of study treatment, participants are followed up at every 3 months for 12 months and then every 6 months for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* ESCLATION COHORT: Patients must have a diagnosis of newly diagnosed and/ or relapsed/refractory AML with any of the following:

  * Confirmed translocation involving 11q23
  * Partial tandem duplication(PTD) of the MLL gene (on 11q23)
  * FLT3-ITD (internal tandem duplication)
  * Increased Fgf2 in serum (2 standard deviations above control serum samples)
  * HOX(A9/A10) over-expression in bone marrow ( 2 standard deviations above control values in CD34+ cells from normal subjects)
  * Note: Relapsed or refractory AML is defined as either:

    * Recurrence of disease after a complete remission (CR), or
    * Failure to achieve CR with initial therapy
* EXPANSION COHORT: Patients must have a diagnosis of newly diagnosed AML with any of the following:

  * Confirmed translocation involving 11q23
  * Partial tandem duplication (PTD) of the MLL gene (on 11q23)
  * FLT3-ITD (internal tandem duplication)
  * Increased Fgf2 in serum (2 standard deviations above control serum samples)
  * HOX(A9/A10) over-expression in bone marrow (2 standard deviations above control values in CD34+ cells from normal subjects)
  * Note: Patients with secondary AML are eligible for enrollment into the trial (in both cohorts); secondary AML is defined as AML that has developed in a person with a history of antecedent blood count abnormalities, or myelodysplastic syndromes (MDS), or a myeloproliferative disorder (excluding chronic myeloid leukemia); or a history of prior chemotherapy or radiation therapy for a disease other than AML
* Patients who are not candidates for, or decline, intensive therapy
* Patients must exhibit an ECOG performance status 0-3
* International normalized ratio (INR) ? 2 (If coagulopathy is related to disease, this criterion does not apply) within14 days prior to registration
* Prothrombin time (PT) and partial thromboplastin time (PTT) ? 1.5 x of institutional upper limit of normal (ULN) (Note: If coagulopathy is related to disease, this criteria do not apply) within14 days prior to registration
* Total bilirubin ? 1.5 x of institutional ULN within14 days prior to registration
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SPGT]) 1.5 X institutional upper limit of normal (ULN) within14 days prior to registration
* Creatinine 2 x ULN OR creatinine clearance > 30 mL/min based on the Cockroft-Gault glomerular filtration rate (GFR) estimation
* Females of child-bearing potential (FOCBP) and males must agree to use medically acceptable method of contraception (e.g. a method which results in a low failure rate of less than 1% per year when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner for participating females, latex condoms for participating males, sexual abstinence) prior to study entry, for the duration of study participation, and for 3 months following completion of therapy; should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; if the female partner of a male participant becomes pregnant he should inform the treating physician and the female partner should contact her treating physician immediately

  * NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* FOCBP must have a negative pregnancy test (beta-human chorionic gonadotropin [HCG] test in urine or serum) within 7 days prior to registration on study (Note: The test will have to be repeated if cycle 1 day1 is more than 3 days from registration)
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study
* Patients must agree/be able to comply with all protocol specific requirements

Exclusion Criteria:

* Patients who have received chemo-, hormone-, radio or immunotherapy or therapy with monoclonal antibodies or small tyrosine kinase inhibitors within the past 14 days prior to start of treatment or those who have not recovered from adverse events attributed to the agent to grade 1 or baseline

  * Exceptions for prior treatments are:

    * Hydroxyurea for increased blast count (no washout period required; it can be continued throughout the first cycle of therapy)
    * Leukapheresis for leukocytosis (no wash out period required; it can be continued during the study)

      * Note: If patient is registered prior to completion of washout, start date of treatment will need to be confirmed prior to registration; please see assigned quality assurance monitor (QAM) with questions
* Patients who have received any other investigational product within14 days of treatment are not eligible for this study; a wash out period ? 14 days or 5 half- lives (whichever is greater) is required from investigational treatment, prior to start of study treatment; please Note:

  * If patient is registered prior to completion of washout, start date of treatment will need to be confirmed prior to registration; please see assigned QAM with questions
  * The ?5 half-lives? time period will be determined by investigational pharmacy
  * If half life is not known and cannot be predicted, then wash out of ? 14 days is required
* Patients who have had major injuries and/or surgery within the past 4 weeks (< 28 days) prior to registration with incomplete wound healing and/or planned surgery while the patient is on study treatment
* Patients who have proteinuria CTCAE version (v)4.03 grade 2 or greater within < 30 days of registration
* Patients who have significant cardiovascular diseases are not eligible; these are:

  * Uncontrolled hypertension
  * Unstable angina
  * History of infarction within the past 12 months prior to start of study treatment
  * Congestive heart failure > New York Heart Association (NYHA) II
  * Serious uncontrolled cardiac arrhythmia
  * Pericardial effusion
* Patients requiring therapeutic anticoagulation with drugs requiring INR monitoring or anti-platelet therapy, except for acetylsalicylic acid (aspirin) ? 325 mg per day, are not eligible
* Patients with acute promyelocytic leukemia (APL) are not eligible
* Patients with known or suspected central nervous system (CNS) leukemia are not eligible
* Patients with known extramedullary leukemia are not eligible
* Patients who have received prior treatment with nintedanib or any other VEGFR inhibitor are not eligible
* Patients with known hypersensitivity to nintedanib or 5-azacitidine or who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to nintedanib or 5-azacitidine are not eligible
* Patients with hypersensitivity to mannitol are not eligible; patients who have known hypersensitivity to peanut or soya, any other trial drug, or their excipients, or to contrast media are not eligible
* Patients with known active or history of chronic hepatitis C and/or B infection, known HIV infection and active alcohol or drug abuse are not eligible.
* Patient with HIV who require anti-viral or supportive care that interacts with the study drugs are not eligible
* Patients must not have a concurrent active malignancy for which they are receiving treatment
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Active uncontrolled infection
  * Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or active ulcers (gastrointestinal tract, skin) or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient?s safety or study endpoints
* Female patients who are pregnant or nursing are not eligible
* Patients who are unable to swallow oral gel capsules are not eligible
* Patients who have gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-11-14 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 28 days
  Will be defined as the highest dose that causes dose limiting toxicities (DLTs) in < 2 of 6 patients.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 24 months
  Adverse event assessments and laboratory tests will be performed at baseline, and continuously throughout the study at the beginning of each subsequent cycle.
Overall survival | Up to 24 months
  Will be summarized using Kaplan-Meier curves. Median overall survival with 95% confidence interval will be calculated.
Complete remission (CR) rate | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Altman, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States